CLINICAL TRIAL: NCT03745170
Title: Efficacy and Safety Evaluation of Sintilimab or Placebo in Combination With XELOX as First Line Treatment in Patients With Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI308E301
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab+ Oxaliplatin +capecitabine (Experimental)
  Interventions: Drug: Sintilimab; Drug: Oxaliplatin; Drug: Capecitabine
- placebo +Oxaliplatin + Capecitabine (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: placebo

INTERVENTIONS:
Drug: Sintilimab — Weight<60Kg: 3mg/kg Q3W Weignt>=60Kg:200 mg Q3W on Day 1 by IV infusion
  Other Names: IBI308
  Arms: Sintilimab+ Oxaliplatin +capecitabine
Drug: Oxaliplatin — 130 mg/m^2 Q3W on Day 1 by IV infusion
Drug: Capecitabine — 1000 mg/m^2 orally according to Body Surface Area (BSA) BID Q3W on Days 1-14
Drug: placebo — Weight<60Kg: 3mg/kg Q3W Weignt>=60Kg:200 mg Q3W on Day 1 by IV infusion
  Arms: placebo +Oxaliplatin + Capecitabine

SUMMARY:
The purpose of this study is to estimate overall survival of Sintilimab+ oxaliplatin + capecitabine and placebo+ oxaliplatin + capecitabine, as first-line treatment of patients with advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically confirmed diagnosis of unresectable locally advanced,recurrent or metastatic gastric or GEJ adenocarcinoma.
2. Male or Female at least 18 years of age
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Did not receive neoadjuvant or adjuvant treatment (chemotherapy,radiotherapy, or both) for their disease within the last 6 months
5. Must agree to provide tumor tissue sample, either from a previous surgeryor biopsy , within 6 months or fresh, prior to the start of treatment in this study and Has a PD-L1 status determined by immunohistochemistry (IHC) at a central laboratory
6. Has measurable or non-measurable (but assessable) disease as defined by RECIST 1.1 as determined by investigator assessment.
7. Has adequate organ function.
8. Expected survival>=12 weeks.
9. Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test at the timing of enrollment.
10. Participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 6 months after the last dose of study medication.

Exclusion Criteria:

1. Suspicious active bleeding or obstruction phenomenon and Has difficulty in swallow tablets and food
2. HER2-positive status
3. Has had previous therapy for unresectable locally advanced, recurrent or metastatic gastric/GEJ cancer
4. Has received prior therapy with a dose of cisplatin>=300 mg/m-^2
5. Has grade ≥ 2 peripheral sensory neuropathy
6. Known DPD enzyme deficiency status (>=grade 3 mucosal toxicity in previous fluorouracil treatment)
7. Has received prior therapy with an anti-programmed death (PD)-1, anti-PD-L1, anti-PD L2 , anti-CD137,anti-CTLA-4 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
8. Is currently participating in and receiving study therapy ,except those in the survival follow up period of an investigational agent study or non-interventional study .
9. Received systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 4 weeks of first dose. Inhaled or topical steroids ,adrenal replacement steroid doses and steroid of prevention allergic reaction of i.v. contrast agent are permitted in the absence of active autoimmune disease.
10. Received a live vaccine within 4 weeks of the first dose of study medication or plan to receive live vaccine during study period.
11. Has had major surgery (craniotomy, thoracotomy or laparotomy) within 4 weeks prior to first dose of study medication, or anticipation of the need for major surgery during the course of study treatment
12. Known symptomatic central nervous system (CNS) metastasis and/or carcinomatous meningitis. Subjects received prior treatment and have stable disease more than 4 weeks from first dose of study medication.
13. Clinical significant ascites, including which can be detected in percussion, had been ever drained or still need to be controlled currently.
14. Bilateral moderate pleural effusion, or a large amount of pleural effusion on one side, or has caused respiratory dysfunction requiring drainage.
15. Bone metastasis with risk of paraplegia.
16. Active, known or suspected autoimmune disease or has a history of the disease within the last 2 years (subjects with vitiligo, psoriasis, alopecia or Grave's disease, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or type I diabetes mellitus only requiring insulin replacement, but not required systemic treatment in the last 2 years, are permitted to enroll) .
17. Known primary immunodeficiency.
18. Known active tuberculosis.
19. Known history of allogeneic organ or allogeneic hemopoietic stem cell transplantation.
20. Known>=grade 3 allergy or hypersensitivity to oxaliplatin,capecitabine or any monoclonal antibodies.
21. Human Immunodeficiency Virus (HIV) infection (HIV antibody positive).
22. Active or poorly controlled severe infection.
23. Symptomatic congestive heart failure (New York Heart Association grade II-IV) or symptomatic, poorly controlled arrhythmia.
24. Poorly controlled arterial hypertension (SBP ≥ 160mmHg or DBP ≥ 100mmHg) with standard treatment .
25. Prior arterial thromboembolism event, including myocardial infarction, unstable angina, stroke and transient ischemic attack, within 6 months of enrollment.
26. Malnutrition requiring intravenous nutrition, subjects with malnutrition correction≥4 weeks are permitted to enroll.
27. Prior deep vein thrombosis, pulmonary embolism or any other severe thromboembolism events (implanted port or catheter caused thrombosis, or superficial vein thrombosis are not considered as severe thromboembolism) within 3 months before enrollment.
28. History of uncontrolled metabolic disorder, non-malignant organ or systemic disease or secondary carcinomatous reaction, with high medical risk and/or uncertainty of life expectancy evaluation.
29. With hepatic encephalopathy, hepatorenal syndrome or hepatic cirrhosis of Child-Pugh grade B or higher.
30. History of intestinal obstruction or the following diseases: inflammatory bowel disease or extensive bowel resection (partial colonic resection or extensive small bowel resection, concomitant with chronic diarrhea), Crohn's disease, ulcerative colitis.
31. Known acute or chronic active hepatitis B infection (positive HBsAg and HBV DNA ≥ 200 IU/mL or ≥ 10^3 copies/mL positive) infection or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive) infection.
32. History of gastrointestinal perforation and /or fistula within 6 months before enrollment.
33. Subjects with interstitial lung disease requiring steroids therapy.
34. Other primary malignancy, with the exception of:

    1. Malignancy which achieved complete response for at least 2 years before enrollment and do not need other treatment during study period;Curative malignancy, without active disease in the last 5 years and with very low recurrence risk;
    2. Non-melanoma skin cancer or malignant freckle-like nevus with adequate treatment and no evidence of recurrence ;
    3. Adequately treated in-situ carcinoma.
35. Women who are pregnant or nursing.
36. Other acute or chronic diseases, mental illness, or abnormal laboratory test results that may lead to the following outcomes: increase the risk of participating in study or study drug administration, or interfere with the interpretation of the study results and considered by investigator as "NOT" eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Approximately 40 months after the first participant is randomized
  Overall survival (OS)of Sintilimab in combination with oxaliplatin + fluoropyrimidine versus placebo+oxaliplatin + fluoropyrimidine in all randomized participants;Overall survival(OS) of Sintilimab + oxaliplatin + capecitabine versus placebo+ oxaliplatin + capecitabine in participants with programmed cell death ligand 1 (PD-L1) expressing tumors (CPS>=10)

SECONDARY OUTCOMES:
Progression Free Survivla (PFS) | Approximately 40 months after the first participant is randomized
  Progression Free Survivla (PFS) of Sintilimab in combination with oxaliplatin + fluoropyrimidine versus placebo+oxaliplatin + fluoropyrimidine in all randomized participants and PD-L1 expression participants(CPS>=10)
Duration of Response (DoR) | Approximately 40 months after the first participant is randomized
  Duration of Response (DoR) of Sintilimab in combination with oxaliplatin + fluoropyrimidine versus placebo+oxaliplatin + fluoropyrimidine in all randomized participants and PD-L1 expression participants(CPS>=10)
Objective Response Rate (ORR) | Approximately 40 months after the first participant is randomized
  Objective Response Rate (ORR) of Sintilimab in combination with oxaliplatin + fluoropyrimidine versus placebo+oxaliplatin + fluoropyrimidine in all randomized participants and PD-L1 expression participants(CPS>=10) per RESIST v1,1
Disease Control Rate (DCR) | Approximately 40 months after the first participant is randomized
  Disease Control Rate (DCR) of Sintilimab + oxaliplatin + capecitabine versus placebo+ oxaliplatin + capecitabine in in all randomized participants . and PD-L1 expression participants(CPS>=10)
Number of participants experiencing clinical and laboratory adverse events (AEs) | Approximately 40 months after the first participant is randomized
  Safety of Sintilimab in combination with oxaliplatin + fluoropyrimidine versus oxaliplatin + fluoropyrimidine in all randomized participants and PD-L1 expression participants(CPS>=10)

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center,Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wu H, Shu W, Ding Y, Li Q, Li N, Wang Q, Chen Y, Han Y, Huang D, Jiang H. The immune signatures predict gastric/gastroesophageal junction cancer response to first-line anti-PD-1 blockade or chemotherapy. BMC Cancer. 2025 Aug 25;25(1):1369. doi: 10.1186/s12885-025-14805-6. PMID 40851062
- [Derived] Li W, Wan L. Cost-utility of sintilimab plus chemotherapy vs chemotherapy as first-line treatment of advanced gastric or gastroesophageal junction cancer in China. Expert Rev Pharmacoecon Outcomes Res. 2024 Jun;24(5):671-678. doi: 10.1080/14737167.2024.2341859. Epub 2024 Apr 11. PMID 38594905
- [Derived] Xu J, Jiang H, Pan Y, Gu K, Cang S, Han L, Shu Y, Li J, Zhao J, Pan H, Luo S, Qin Y, Guo Q, Bai Y, Ling Y, Yang J, Yan Z, Yang L, Tang Y, He Y, Zhang L, Liang X, Niu Z, Zhang J, Mao Y, Guo Y, Peng B, Li Z, Liu Y, Wang Y, Zhou H; ORIENT-16 Investigators. Sintilimab Plus Chemotherapy for Unresectable Gastric or Gastroesophageal Junction Cancer: The ORIENT-16 Randomized Clinical Trial. JAMA. 2023 Dec 5;330(21):2064-2074. doi: 10.1001/jama.2023.19918. PMID 38051328